CLINICAL TRIAL: NCT06165718
Title: A Multicenter, Observational Study for the Clinical Roadmap and Prognosis of Pulmonary Artery Sarcoma.
Brief Title: Study for the Clinical Roadmap and Prognosis of Pulmonary Artery Sarcoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Beijing Chao Yang Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Sir Run Run Shaw Hospital (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Wanmu Xie, Professor, China-Japan Friendship Hospital
Other Study IDs: Roadmap for PAS-2022
Record Dates: First submitted 2023-12-04; First posted 2023-12-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Artery Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study in which patients with pulmonary artery sarcoma were followed up for at least 36 months and survival was investigated.

DETAILED DESCRIPTION:
This is an observational study covering mainland China, and patients with pulmonary artery sarcoma were followed up for at least 36 months and survival was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography pulmonary angiography indicated that there were intraluminal defects
* Malignant histopathology was sarcoma
* Informed consent form was signed

Exclusion Criteria:

* Life expectancy was less than 3 months due to diseases other than pulmonary artery sarcoma
* Expected inability to complete follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonary artery sarcoma patients expected to complete follow-up
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36 months
  Time to death or disease progression

SECONDARY OUTCOMES:
Overall survival | 36 months
  Time to death
Postoperative survival | 36 months
  Time from surgery to death

CONTACTS AND LOCATIONS:
Overall Officials: Wanmu Xie, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China